CLINICAL TRIAL: NCT02536404
Title: Extension Study of APD334-003 in Patients With Moderately to Severely Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: APD334-005
Record Dates: First submitted 2015-08-24; First posted 2015-08-31 (Estimated); Results first posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrasimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etrasimod 2 mg (Experimental)
  Interventions: Drug: Etrasimod
- Placebo (Active Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etrasimod
  Other Names: APD334
  Arms: Etrasimod 2 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether etrasimod (APD334) is a safe and effective treatment for ulcerative colitis after 52 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants who completed the APD334-003 (NCT02447302) study

Exclusion Criteria:

* Participants who did not complete the APD334-003 study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arena CT.gov Administrator, Study Director — Arena Pharmaceuticals
Locations (127):
- United States (31):
  - Arena 1119, Birmingham, Alabama
  - Arena 1133, Dothan, Alabama
  - Arena 1143, Thousand Oaks, California
  - Arena 1107, Hollywood, Florida
  - Arena 1138, Miami, Florida
  - Arena 1123, Naples, Florida
  - Arena 1141, Orlando, Florida
  - Arena 1106, Port Orange, Florida
  - Arena 1137, Sweetwater, Florida
  - Arena 1131, Chicago, Illinois
  - Arena 1139, Hoffman Estates, Illinois
  - Arena 1127, Urbana, Illinois
  - Arena 1113, Chevy Chase, Maryland
  - Arena 1142, Traverse City, Michigan
  - Arena 1111, Troy, Michigan
  - Arena 1109, Great Neck, New York
  - Arena 1114, Rochester, New York
  - Arena 1118, Raleigh, North Carolina
  - Arena 1112, Cincinnati, Ohio
  - Arena 1117, Pittsburgh, Pennsylvania
  - Arena 1105, Germantown, Tennessee
  - Arena 1102, Hermitage, Tennessee
  - Arena 1136, DeSoto, Texas
  - Arena 1121, Houston, Texas
  - Arena 1116, Temple, Texas
  - Arena 1103, Ogden, Utah
  - Arena 1130, Richmond, Virginia
  - Arena 1128, Roanoke, Virginia
  - Arena 1115, Seattle, Washington
  - Arena 1101, Seattle, Washington
  - Arena 1108, Wauwatosa, Wisconsin
- Australia (3):
  - Arena 1604, Kingswood
  - Arena 1605, Randwick
  - Arena 1607, Subiaco
- Arena 1490, Vienna, Austria
- Belgium (3):
  - Arena 1472, Edegem
  - Arena 1464, Kortrijk
  - Arena 1473, Leuven
- Bulgaria (6):
  - Arena 1421, Rousse
  - Arena 1417, Sofia
  - Arena 1410, Sofia
  - Arena 1409, Sofia
  - Arena 1407, Sofia
  - Arena 1425, Varna
- Canada (6):
  - Arena 1202, Winnipeg, Manitoba
  - Arena 1210, Bridgewater, Nova Scotia
  - Arena 1208, Greater Sudbury, Ontario
  - Arena 1209, Greater Sudbury, Ontario
  - Arena 1206, London, Ontario
  - Arena 1204, Toronto, Ontario
- Arena 1455, Prague, Czechia
- France (7):
  - Arena 1443, Amiens
  - Arena 1418, Clichy
  - Arena 1437, Lille
  - Arena 1476, Paris
  - Arena 1480, Pierre-Bénite
  - Arena 1423, Saint-Etienne
  - Arena 1457, Vandœuvre-lès-Nancy
- Germany (7):
  - Arena 1479, Hamburg
  - Arena 1422, Hamburg
  - Arena 1470, Hanover
  - Arena 1446, Kiel
  - Arena 1489, Leipzig
  - Arena 1497, Oldenburg
  - Arena 1444, Ulm
- Hungary (7):
  - Arena 1478, Békéscsaba
  - Arena 1431, Budapest
  - Arena 1471, Budapest
  - Arena 1492, Budapest
  - Arena 1505, Debrecen
  - Arena 1474, Debrecen
  - Arena 1477, Szombathely
- Israel (5):
  - Arena 1705, Beersheba
  - Arena 1702, Haifa
  - Arena 1706, Holon
  - Arena 1704, Jerusalem
  - Arena 1703, Petah Tikva
- Latvia (2):
  - Arena 1462, Riga
  - Arena 1475, Riga
- Arena 1484, Vilnius, Lithuania
- Arena 1601, Christchurch, New Zealand
- Poland (9):
  - Arena 1439, Bydgoszcz
  - Arena 1486, Elblag
  - Arena 1495, Kielce
  - Arena 1451, Krakow
  - Arena 1438, Lodz
  - Arena 1458, Poznan
  - Arena 1428, Rzeszów
  - Arena 1456, Sopot
  - Arena 1494, Wroclaw
- Romania (7):
  - Arena 1491, Bucharest
  - Arena 1406, Bucharest
  - Arena 1441, Bucharest
  - Arena 1436, Iași
  - Arena 1420, Oradea
  - Arena 1405, Timișoara
  - Arena 1493, Timișoara
- Russia (6):
  - Arena 1500, Krasnoyarsk
  - Arena 1504, Novosibirsk
  - Arena 1419, Rostov-on-Don
  - Arena 1498, Saint Petersburg
  - Arena 1448, Saint Petersburg
  - Arena 1465, Samara
- South Korea (3):
  - Arena 1615, Wŏnju, Gangwon-do
  - Arena 1614, Daegu
  - Arena 1610, Incheon
- Spain (6):
  - Arena 1403, Barcelona
  - Arena 1460, Barcelona
  - Arena 1481, Madrid
  - Arena 1430, Pontevedra
  - Arena 1432, Santiago de Compostela
  - Arena 1469, Seville
- Ukraine (12):
  - Arena 1424, Chernivtsi
  - Arena 1445, Ivano-Frankivsk
  - Arena 1454, Kharkiv
  - Arena 1459, Kharkiv
  - Arena 1466, Kiev
  - Arena 1411, Kiev
  - Arena 1408, Kyiv
  - Arena 1506, Kyiv
  - Arena 1414, Odesa
  - Arena 1433, Uzhhorod
  - Arena 1416, Vinnytsia
  - Arena 1501, Vinnytsia
- United Kingdom (3):
  - Arena 1302, London
  - Arena 1304, Torquay
  - Arena 1303, Wolverhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vermeire S, Rubin DT, Peyrin-Biroulet L, Dubinsky MC, Regueiro M, Irving PM, Goetsch M, Lazin K, Gu G, Wu J, Modesto I, McDonnell A, Guo X, Green J, Dalam AB, Yarur AJ. Cardiovascular events observed among patients in the etrasimod clinical programme: an integrated safety analysis of patients with moderately to severely active ulcerative colitis. BMJ Open Gastroenterol. 2025 Jan 8;12(1):e001516. doi: 10.1136/bmjgast-2024-001516. PMID 39778975

RESULTS

PARTICIPANT FLOW:
Groups:
- Etrasimod 2 mg: Participants received etrasimod 2 milligrams (mg) tablet by mouth, once daily for 34 weeks in fasted state.
- Placebo: Participants received matching placebo tablet by mouth, once daily for 34 weeks in fasted state.
Period: Overall Study
Arm/Group | Etrasimod 2 mg | Placebo
Started | 112 | 6
Completed | 92 | 5
Not Completed | 20 | 1
Not completed — Adverse Event | 5 | 0
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Physician Decision | 10 | 0
Not completed — Sponsor decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for members of the Safety Population, comprised of all participants who received study medication in the extension study APD334-005 (NCT02536404).
Groups:
- Total: Total of all reporting groups
Arm/Group | Etrasimod 2 mg | Placebo | Total
Number analyzed (Participants) | 112 | 6 | 118
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (13.25) | 50.2 (13.93) | 44.0 (13.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 3 | 47
  Male | 68 | 3 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 108 | 6 | 114
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 104 | 6 | 110
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (SAEs)
Description: A TEAE was defined as any adverse event (AE) that occurred after the first dose of study drug in the APD334-005 (NCT02536404) study, including any AE that started in Study APD334-003 (NCT02447302) and was ongoing, worsened, or ended in Study APD334-005. A SAE was any untoward medical occurrence that at any dose resulted in the following outcomes: death, was life-threatening, required/prolonged hospitalization, disability/incapacity, congenital anomaly/birth defect, and important medical events.
Time Frame: Up to Week 48 (up to 30 days following discontinuation of the study drug)
Population: Safety Population: All randomized participants who received study medication in the extension study APD334-005
Measure: Count of Participants; unit: Participants
Groups:
- Etrasimod 2 mg: Participants received etrasimod 2 mg tablet by mouth, once daily for 34 weeks in fasted state.
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 112 | 6
Participants
  TEAEs | 67 | 5
  Treatment-emergent SAEs | 7 | 0

2. Secondary Outcome: Proportion of Participants Who Achieved Clinical Response
Description: A participant was considered to have achieved clinical response if he/she met the criteria of clinical remission or met criteria of clinical response. Clinical remission was defined as individual subscores of the 3-component Mayo Clinic score as follows: (1) an endoscopy score (using flexible proctosigmoidoscopy) of 0 or 1, (2) a rectal bleeding score of 0, and (3) a stool frequency score of 0 or 1 with a decrease of ≥ 1 point at Week 46 compared to APD334-003 baseline. Clinical response was defined as a decrease in 3-component Mayo Clinic score of ≥ 2 points and at least 30% with either a decrease of rectal bleeding of ≥ 1 or rectal bleeding score of 0 or 1 at Week 46 compared with baseline of study APD334-003. A score of 0 = normal and 1 = mild disease.
Time Frame: Week 46 (extension study APD334-005)
Population: Completers Population Evaluable Cohort: All participants who received at least 1 dose of etrasimod or placebo and completed the extension study APD334-005
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 84 | 4
Percentage of participants | 78.6 [69.9 to 85.7] | 75.0 [24.9 to 98.7]

3. Secondary Outcome: Proportion of Participants Who Achieved Clinical Response at Week 12 in APD334-003 and Maintained Clinical Response at Week 46 in APD334-005
Description: as for outcome 2
Time Frame: Week 12 (core study APD334-003) and Week 46 (extension study APD334-005)
Population: Completers Population Evaluable Cohort
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 84 | 4
Percentage of participants | 39.3 [30.3 to 48.8] | 50.0 [9.8 to 90.2]

4. Secondary Outcome: Proportion of Participants Who Achieved Clinical Remission
Description: A participant was considered to have achieved clinical remission if he/she had: (1) an endoscopy score (using flexible proctosigmoidoscopy) of 0 or 1, (2) a rectal bleeding score of 0, and (3) a stool frequency score of 0 or 1 with a decrease of ≥ 1 point at Week 46 compared with baseline of study APD334-003. A score of 0 = normal and 1 = mild disease.
Time Frame: Week 46 (extension study APD334-005)
Population: Completers Population Evaluable Cohort
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 84 | 4
Percentage of participants | 39.3 [30.3 to 48.8] | 25.0 [1.3 to 75.1]

5. Secondary Outcome: Proportion of Participants Who Achieved Clinical Remission at Week 12 in APD334-003 and Also Maintained Clinical Remission at Week 46 in APD334-005
Description: as for outcome 4
Time Frame: Week 12 (core study APD334-003) and Week 46 (extension study APD334-005)
Population: Completers Population Evaluable Cohort
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 84 | 4
Percentage of participants | 14.3 [8.5 to 22.1] | 0 [0.0 to 52.7]

ADVERSE EVENTS:
Time Frame: Up to Week 48 (up to 30 days following discontinuation of the study drug)
Description: A TEAE was defined as any adverse event (AE) that occurred after the first dose of study drug in the APD334-005 (NCT02536404) study, including any AE that started in Study APD334-003 (NCT02447302) and was ongoing, worsened, or ended in Study APD334-005. A SAE was any untoward medical occurrence that at any dose resulted in the following outcomes: death, was life-threatening, required/prolonged hospitalization, disability/incapacity, congenital anomaly/birth defect, and important medical events.
Arm/Group | Etrasimod 2 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/6
Serious Adverse Events (participants affected / at risk) | 7/112 | 0/6
Other Adverse Events (participants affected / at risk) | 66/112 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etrasimod 2 mg (N=112) | Placebo (N=6)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 3 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Proctitis ulcerative (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Fine motor skill dysfunction (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etrasimod 2 mg (N=112) | Placebo (N=6)
Gamma-glutamyltransferase increased (Investigations) | 10 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Faecal calprotectin increased (Investigations) | 3 | 1
Hepatic enzyme increased (Investigations) | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 10 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Headache (Nervous system disorders) | 5 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1
Vitreous (Eye disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 16 | 1
Nausea (Gastrointestinal disorders) | 5 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Premenstrual headache (Reproductive system and breast disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 6 | 2
Upper respiratory tract infection (Infections and infestations) | 7 | 0
Gastroenteritis (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 1
Tooth infection (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT02536404/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT02536404/SAP_001.pdf